CLINICAL TRIAL: NCT00514605
Title: A Study to Evaluate the Point-of-Care Use and Laboratory Investigational Testing of INSTI™ HIV-1 Antibody Test Kit in Volunteer Subjects at Risk for HIV Infection
Brief Title: Testing of INSTI™ HIV-1 Antibody Test Kit in Volunteer Subjects at Risk for HIV Infection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: bioLytical Laboratories (Industry)
Responsible Party: Rick Galli, Biolytical Laboratories
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2007-01
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: HIV Infections
Keywords: HIV 1; AIDS; Assay; Rapid Test; HIV-1; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Behavioral counseling — Standard-of-Care counseling at the Point-of-Care.
Device: HIV-1 Antibody Test Kit — Assay to detect HIV antibodies
  Other Names: INSTI™ HIV-1 Antibody Test Kit

SUMMARY:
Each year up to 22 million persons in the US are tested for HIV. Currently available "rapid" tests do not provide test results for at least 30 minutes from the collection of serum and plasma from the subject. Providing accurate test results in less than a minute would make it easier to make timely decisions about treatment and counselling.

This study will compare results of an experimental rapid test to existing standards to determine if the test can reliably and accurately diagnose HIV in less than one minute.

DETAILED DESCRIPTION:
The primary objective is to determine if INSTI™ performed with finger-stick whole blood, venous whole blood, and plasma demonstrates at least 98.0% sensitivity and specificity compared to an FDA-approved HIV testing algorithm.

The study will have two parts. The first part of the study will be conducted in institutions where HIV testing is routinely performed and where HIV counseling is offered [i.e. point of care (POC) centers]. The second part of the study will be conducted in a central laboratory that routinely conducts laboratory-based HIV testing using an FDA-licensed HIV-1 ELISA and Western blot test.

Geographically diverse POCs will be selected in the USA. Approximately 15-20 POCs are planned. Approximately 2,500 subjects will participate in the study including 1,500 subjects with unknown HIV status and 1,000 seropositive subjects. Across these POC sites, voluntary testing of 1500 subjects with unknown HIV status is planned with at least 500 of these subjects being high risk. Samples will be obtained from consenting subjects in the voluntary testing population including high-risk and known HIV 1 seropositive individuals.

Each subject is to receive an INSTI™ on finger-stick blood and parallel HIV testing of EDTA-treated venous whole blood and plasma samples will be conducted at a central laboratory.

The results of INSTI™ will not be given to the subject. The subject will be given the results of the POC HIV test only, per their standard of care procedures. Subsequent subject care decisions will NOT be based on the results of INSTI™.

ELIGIBILITY:
Inclusion Criteria:

* Unknown HIV status who are undergoing voluntary testing for HIV infection in a POC clinic setting or known HIV seropositive subjects willing to be re-tested.
* Ability to give proper informed consent, or have legal parent or guardian provide consent.
* Willingness to participate in a POC standard of care HIV counseling and testing program and receive POC standard of care test results
* Willingness to provide the necessary volume of whole blood collected through venous blood draw and finger stick (approximately 10 ml)

Exclusion Criteria:

* Subject self-report of history of multiple myeloma
* Subject self-report of history of long-term anti-retroviral therapy with known low or non-existent antibody titre (sero-inversion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2007-07; Primary Completion 2007-11-20 (Actual); Study Completion 2007-11-20 (Actual)

PRIMARY OUTCOMES:
INSTI™ performed with finger-stick whole blood, venous whole blood, and plasma demonstrates at least 98.0% sensitivity and specificity compared to an FDA-approved HIV testing algorithm | <1 week

SECONDARY OUTCOMES:
The percentage of INSTI™ results that agree between finger-stick whole blood, venous whole blood, and plasma. | < 1 week

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - LA County STD Program, Los Angeles, California
  - Michael Sumero, MD, Palm Springs, California
  - UCSD Antiviral Research Center, San Diego, California
  - Denver Public Health, Denver, Colorado
  - Midland Medical, Fort Lauderdale, Florida
  - University of Maryland, Baltimore School of Medicine, Baltimore, Maryland
  - Department of Epidemiology, Johns Hopkins School of Public Health, Baltimore, Maryland
  - Crossroads Clinic, Jackson, Mississippi
  - National Development and Research Institute, New York, New York
  - New York Academy of Medicine, New York, New York
  - Mazzoni Center, Philadelphia, Pennsylvania
  - AIDS/HIV Services Group, Charlottesville, Virginia
  - Richmond AIDS Consortium, Richmond, Virginia
  - Cross Over Ministry, Richmond, Virginia